CLINICAL TRIAL: NCT01328353
Title: Telehealth Nursing Intervention for Children With Complex Health Care Needs
Brief Title: Telehealth Nursing Intervention for Children With Complex Health Care Needs (CCHCN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0908M70627
Record Dates: First submitted 2011-03-25; First posted 2011-04-04 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Unplanned Use of Health Care Services
Keywords: triage; aprn; telehealth; CCHCN; advanced practice nurse; improve family quality of life; reduce unplanned use of health care services; telehealth triage intervention
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control group (No Intervention): Control group arm follows usual care
- Intervention group arm 1 (Experimental): Intervention group arm 1 receives aprn/telephone care coordination
  Interventions: Other: telehealth plus aprn triage
- Intervention group arm 2 (Experimental): Intervention group arm 2 receives aprn/telephone/video care coordination
  Interventions: Other: telehealth plus aprn triage

INTERVENTIONS:
Other: telehealth plus aprn triage — aprn using either telephone or telephone plus video conferencing will provide triage for CCHCN
  Other Names: APRN
  Arms: Intervention group arm 1; Intervention group arm 2

SUMMARY:
The overall objective of this study is to evaluate the effectiveness of a telehealth care coordination and case management nursing intervention for children with complex special health care needs.

DETAILED DESCRIPTION:
Children with complex special health care needs are those children who have multiple, complex, chronic health conditions who require health and related services of a type or amount beyond that required by children generally. When these children are hospitalized, they receive services as part of an integrated system that provides centralized record keeping and care orders, clearly identified roles and methods of communication for health professionals involved in their care, an established method to obtain equipment and supplies, and regular monitoring of the child's condition. However, when the same child is cared for at home, services are often fragmented, and rarely accessed and delivered in a coordinated system. The task of coordinating services and sharing information between providers almost always becomes the responsibility of the parent or guardian. Families report that their greatest challenges are the stress of coordinating multiple providers, and the disconnect and lack of communication between services and providers. This study will address these issues, using an advanced practice nurse (APN) program of telehealth care coordination and case management in support of these families. Either the telephone or telephone plus interactive video are used by an advanced practice nurse to provide care coordination and case management. Goals of the program are to (1) reduce the number of crisis or unplanned uses of health care services and increase the number of non-crisis or planned health care service usage, (2) improve the QL (quality of life) for these children and their families, and (3) reduce the deficit between help needed and help received for the families in caring for these children. The study objective will be accomplished using a three armed randomized controlled trial. Children will be randomized into a control group receiving usual care that includes LPN (Licensed practical nurse)-delivered care coordination and RN (registered nurse)-delivered telephone triage, an intervention group receiving APN-delivered telephone care coordination and case management, and another intervention group receiving APN-delivered telephone + video care coordination and case management services. It is hypothesized that as the level of telehealth use in coordination and management increases the utilization of unplanned, or crisis, health care service utilization will decrease, that families will receive more of their needed care, and quality of life for the children and their families will improve

ELIGIBILITY:
Inclusion Criteria:

* Children with complex health care needs, in the patient population of the Special Needs Clinic, St Paul Children's Hospital

Exclusion Criteria:

* Healthy children
* CCHCN children not seen in the Special Needs Clinic at St Paul Children's Hospital

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the number of crisis or unplanned uses of health care services by enrolled subject, based on data collected in the Health Care Service Utilization calendar maintained by study subjects, and from the subjects' EMR | 2 year RCT follow-up
  This measure will show if the intervention can shift the number of crisis and unplanned health care services utilized to planned service utilization, based on data collected from the subjects' Health Care Service Utilization calendars and their EMR

SECONDARY OUTCOMES:
To measure changes in quality of life for CCHCN and their families over the study period, using scores from the PedsQL and PedsQL Family Impact Module instruments. | 2 years RCT follow-up
  These measures will determine the effectiveness of the intervention on improving the quality of life for CCHCN subjects and their families, based on scores from the Peds QL and PedsQL Family Module survey instruments
To measure the deficit between help needed and help received using the Discrepancy Visual Analog scale | 2 years RCT follow-up
  To measure the effectiveness of the intervention on reducing the discrepancy between parents' reported need for help from others and their reported receipt of help from others using the Discrepancy Visual Analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Finkelstein, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Univ Minnesota and St Paul Childrens Hospital and Clinic, Minneapolis, Minnesota, United States